CLINICAL TRIAL: NCT01266187
Title: Perioperative Chemotherapy With FOLFOX Plus Cetuximab Versus Adjuvant FOLFOX Plus Cetuximab for Patients With Resectable Liver Metastases of Colorectal Carcinoma
Brief Title: Treatment Regimens for Patients With Resectable Liver Metastases (PANTER Study)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulities
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTC-A10-005
Record Dates: First submitted 2010-12-20; First posted 2010-12-24 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Liver Metastasis
Keywords: FOLFOX; liver metastasis; cetuximab
MeSH Terms: interventions — Folfox protocol; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm B (Experimental): 12 weeks FOLFOX + cetuximab -> 4 weeks rest -> surgery
  -> 4-8 weeks rest -> 12 weeks FOLFOX + cetuximab
  Interventions: Procedure: perioperative/Folfox + cetuximab
- Arm A (Active Comparator): surgery -> 4-8 weeks rest -> 24 weeks FOLFOX + cetuximab
  Interventions: Procedure: adjuvant surgery + FOLFOX + cetuximab

INTERVENTIONS:
Procedure: adjuvant surgery + FOLFOX + cetuximab — surgery -> 4-8 weeks rest -> 24 weeks FOLFOX + cetuximab
  Arms: Arm A
Procedure: perioperative/Folfox + cetuximab — 12 weeks FOLFOX + cetuximab -> 4 weeks rest -> surgery
  -> 4-8 weeks rest -> 12 weeks FOLFOX + cetuximab
  Arms: Arm B

SUMMARY:
Is a perioperative chemotherapy based on FOLFOX and Cetuximab (K-RAS wild-type) associated with a higher rate of postoperative complications in patients with resectable colorectal liver metastases as compared to only adjuvant FOLFOX and chemotherapy? Are there any differences for disease free survival between periand postoperative treatment in patients with >3 liver metastases or at least one metastasis > or = 5 cm in diameter?

DETAILED DESCRIPTION:
In recent years chemotherapy based on FOLFOX and cetuximab has become a standard treatment in patients with colorectal liver metastases. Recently, the analysis of the CELIM trial reported response rates of 70% in patients with initially unresectable colorectal liver metastases treated with FOLFOX + Cetuximab. 46% of the patients had their metastases R0 or R1 resected or a ablation by radiofrequency with an overall 34% R0 resection rate. In recent studies, adjuvant chemotherapy with FOLFOX leads to a prolongation of disease free survival after successful resection of colorectal liver metastases, but there is not sufficient data concerning a perioperative regimen. In only one study of Nordlinger et al. a trend in progression-free survival could be reached in patients receiving a perioperative FOLFOX-therapy, but without reaching statistical significance. Furthermore those patients displayed a significantly higher rate of postoperative complications and morbidity. Although the advantages of perioperative treatment are not proven, this concept has become more and more popular in recent years, mainly because of a lack of guidelines. Thus the aim of our study is to compare the complication rate of both therapeutical concepts. Furthermore, secondary objectives (disease-free survival, overall survival, resection rates, response rates, toxicities and quality of life) will be used to estimate the efficacy, feasibility, and safety of both regimens. Perioperative treatment probably has a better efficacy in patients with high tumor burden (>3 liver metastases or one metastasis > or = 5 cm in diameter) with effect on disease free survival and will be investigated in a subgroup analysis.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent obtained prior to any study-specific procedure.
* Age > 18 years
* Proven K-RAS wildtype in primary tumour or metastasis tissue
* Diagnosis of resectable metachronous metastases after complete resection (R0) of primary tumour without gross or microscopic evidence of residual disease. or Diagnosis of resectable synchronous metastases after complete resection (R0) of primary tumour more than 1 month before study or Diagnosis of resectable synchronous metastases with sufficient evidence (i.e., CT scan or diagnostic laparoscopy) that both the primary tumour and liver metastases can be completely resected during the same procedure and resection of primary can be delayed 3-4 months.
* Negative pregnancy test
* Highly effective contraception during treatment and for at least 3 months thereafter in women (defined as pearl index < 1) and men, if the risk of conception exists
* Planned start of study medication between 0 and 3 weeks post randomization
* ECOG performance status 0 or 1 (Appendix 1)
* Adequate hematology: neutrophils > 1,5 /nl, platelets > 100/nl, INR < 1,5, aPTT < 1,5 x UNL
* Adequate biochemistry: total bilirubin < 1,5 x UNL, ASAT and ALAT < 5 x UNL, alkaline phosphatase < 5 x UNL, serum creatinine < 1,5, x UNL.

Exclusion Criteria:

* Patients with any relationship of dependence to the sponsor or the investigator
* Patients committed to an institution (court-ordered or by official orders)
* Extrahepatic metastatic disease
* Proven K-RAS mutation or unknown K-RAS mutational status in tumour tissue
* Oxaliplatin-based adjuvant chemotherapy within 1 year before randomization
* Neuropathy > or = grade 3 (NCI-CTC V4.0) during prior oxaliplatin-based chemotherapy
* Any prior chemotherapy for metastatic disease
* Previous treatment with EGFR antibodies
* Prior non-colorectal malignancies, except adequately treated basalioma of the skin or carcinoma in situ of the cervix.
* Bleeding diathesis or coagulation disorders
* Females with a positive pregnancy test (within 14 days before treatment start) or breast feeding
* Fertile women (<2 years after last menstruation) and women of childbearing potential not willing to use effective means of contraception
* History of psychiatric disability judged by the investigator to be clinically significant, precluding informed consent or interfering with compliance for drug intake
* Clinically significant (i.e. active) cardiovascular disease, e.g. cerebrovascular accidents (<6 months prior to randomization), myocardial infarction (<1 year prior to randomization), Congestive heart failure (NYHA Grades III or IV), uncontrolled hypertension while receiving chronic medication, unstable angina pectoris, significant arrhythmia
* Known peripheral neuropathy, including oxaliplatininduced

  > or = grade 1 (NCI-CTC V4.0). Absence of deep tendon reflexes being the sole neurologicl abnormality does not render the patient ineligible
* Known DPD-deficiency (Dihydropyrimidinedehydrogenase)
* Organ allografts requiring immunosuppressive therapy
* Serious, non-healing wound, ulcer or bone fracture
* Serious intercurrent infections (uncontrolled or requiring treatment)
* Current or recent (within 28 days prior to randomisation) treatment with another investigational drug or participation in another investigational study
* Any contraindications against study medication (including auxiliary substances)
* Patients unwilling to consent the saving and propagation of pseudonymized medical data for study reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Clavien score (> grade 1) | 1 year
  The first primary objective of the study is to compare the postoperative complication rate according to Clavien score (> grade 1) of a perioperative chemotherapy with a postoperative regimen
Disease free survival | 1 year
  A second primary objective of the study is to compare for the patient subgroup with >3 liver metastases or at least one metastasis > or = 5 cm in diameter the median disease free survival.

SECONDARY OUTCOMES:
Secondary objectives | 5 years
  Secondary Objectives:
  * To compare the overall disease-free survival.
  * To compare the overall survival.
  * To compare operation, resection and R0 rates.
  * To compare the safety and chemotherapy-associated toxicity (NCI-CTC V4.0)
  * To compare the effect of a perioperative therapy on healthrelated quality of life (EORTC QLQ-C30 + QLQ-LMC21).
  * To compare the number of cycles, dose intensity and dose modifications applied.
  * To evaluate the response rate (RECIST V1.1 no confirmation of response needed) after preoperative chemotherapy.
  * Resected liver mass

CONTACTS AND LOCATIONS:
Overall Officials: Ulf P Neumann, Prof., Study Director — RWTH Aachen University Hospital
Locations (1):
- Department of Surgery, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany